CLINICAL TRIAL: NCT00508391
Title: Clinical Investigation to Study Safety and Efficacy of the Interventricular Delay Feature of the Lumax HF-T Device for Heart Failure.
Brief Title: Interventricular Delay of Lumax HF-T for Heart Failure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biotronik, Inc. (Industry)
Responsible Party: Clay Cohorn, Clinical Studies Engineer II, Biotronik, Inc.
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: G070019
Record Dates: First submitted 2007-07-26; First posted 2007-07-30 (Estimated); Results first posted 2010-01-18 (Estimated); Last update posted 2010-01-26 (Estimated); Status verified 2010-01

CONDITIONS: Congestive Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Simultaneous 1st, Optimized 2nd (Experimental): Lumax HF-T device programmed to simultaneous biventricular pacing first for 30 days, followed by optimized biventricular pacing for 30 days.
  Interventions: Device: Optimized interventricular delay biventricular pacing
- Optimized 1st, Simultaneous 2nd (Experimental): Lumax HF-T device programmed to optimized biventricular pacing first for 30 days, followed by simultaneous biventricular pacing for 30 days.
  Interventions: Device: Optimized interventricular delay biventricular pacing

INTERVENTIONS:
Device: Optimized interventricular delay biventricular pacing — Lumax HF-T with optimized interventricular delay biventricular pacing
  Other Names: Optimized CRT, Interventricular delay

SUMMARY:
The purpose of this study is to demonstrate that the safety and efficacy of the Lumax HF-T with optimized interventricular delay biventricular pacing (OPT) is non-inferior to the Lumax HF-T with simultaneous biventricular pacing (SIM) in patients with heart failure requiring cardiac resynchronization therapy.

DETAILED DESCRIPTION:
This study is a randomized, double-blinded, crossover, multi-center, prospective trial. The study will consist of up to 122 subjects who require treatment of advanced heart failure through cardiac resynchronization therapy (CRT) with back-up defibrillation capabilities. Eligible patients will have a successfully implanted BIOTRONIK Lumax HF-T CRT-D system and have received simultaneous biventricular pacing for a minimum of 90 days prior to enrollment. The 90-day period is being required to allow the treatment effect of CRT therapy with SIM to be complete and to ensure the patient is receiving a stable and optimal CHF medical regimen. The patients will have the interventricular delay feature programmed after a standardized optimization procedure. Patients, along with study personnel evaluating the study endpoint measures, will be blinded to the type of CRT therapy delivered during the study follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Meet the indications for therapy
* Successfully implanted with a BIOTRONIK Lumax HF-T CRT-D system and have received SIM for a minimum of 30 days prior to enrollment. A successful implantation is defined as having a measured LV pacing threshold which allows for a minimum 1-volt safety margin without any phrenic nerve stimulation at the time of enrollment.
* Treated with stable and optimal CHF medications, which includes an ACE inhibitor (ACE-I) or Angiotensin Receptor Blocker (ARB) at therapeutic dose for 1 month prior to enrollment, if tolerated, and a Beta Blocker that is approved and indicated for HF for 3 months prior to enrollment, if tolerated, with a stable dosage for 1 month prior to enrollment. If the patient is intolerant of ACE-I or beta blockers, documented evidence must be available. Eplerenone requires dosage stability for 1 month prior to enrollment. Diuretics may be used as necessary to keep the patient euvolemic. Therapeutic equivalence for ACE-I substitutions is allowed within the enrollment stability timeliness. Stable is defined as no more than a 100% increase or a 50% decrease in dose.
* Age ≥ 18 years
* Able to understand the nature of the study and give informed consent
* Able to complete all testing required by the clinical protocol, including the 6-minute walk test and QOL questionnaire
* Available for follow-up visits on a regular basis at the investigational site

Exclusion Criteria:

* Meet one or more of the contraindications
* Have a life expectancy of less than 6 months
* Expected to receive heart transplantation within 6 months
* Have had more than 1 CHF-related hospitalization within past 30 days
* Currently receiving IV inotropic medications
* Chronic atrial fibrillation
* Enrolled in another cardiovascular or pharmacological clinical investigation, except for FDA required post-market registries
* Any condition preventing the patient from being able to perform required testing
* Presence of another life-threatening, underlying illness separate from their cardiac disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2007-07; Primary Completion 2008-12 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (19):
- United States (18):
  - Solano Cardiology, Fairfield, California
  - Cardiac Arrhythmia Associates, La Jolla, California
  - Sansum Clinic, Santa Barbara, California
  - Cardiology Associates Medical Group, Ventura, California
  - Cardiac Disease Specialists, P.C., Atlanta, Georgia
  - Georgia Arrhythmia Consultants, Macon, Georgia
  - Fananapazir, Cumberland, Maryland
  - St. Elizabeth's Medical Center, Boston, Massachusetts
  - Michigan Cardiovascular Institute, Saginaw, Michigan
  - SSM Medical Group, St Louis, Missouri
  - Gateway Cardiology, St Louis, Missouri
  - Salem Cardiology, Salem, Oregon
  - Palmetto Cardiology, Columbia, South Carolina
  - Pee Dee Cardiology, Florence, South Carolina
  - Cardiology Consultants, Spartanburg, South Carolina
  - Lone Star Heart Center, Amarillo, Texas
  - Cardiac Associates of Dallas, Dallas, Texas
  - Yakima Heart Center, Yakima, Washington
- University Hospital Zurich, Zurich, Switzerland, Switzerland

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from each investigator's general patient population at the medical clinic and selected according to the study inclusion/exclusion criteria.
Pre-assignment Details: All subjects enrolled in the study were previously implanted with a Lumax HF-T heart failure device. The study utilized an intention-to-treat analysis where subjects were analyzed according to the randomized treatment order, regardless of whether they received the treatment in the order stipulated by the protocol.
Period: First Treatment
Arm/Group | Simultaneous 1st, Optimized 2nd | Optimized 1st, Simultaneous 2nd
Started | 60 | 62
Completed | 54 | 59
Not Completed | 6 | 3
Not completed — Withdrawal by Subject | 6 | 3
Period: Second Treatment
Arm/Group | Simultaneous 1st, Optimized 2nd | Optimized 1st, Simultaneous 2nd
Started | 54 | 59
Completed | 52 | 59
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Simultaneous 1st, Optimized 2nd | Optimized 1st, Simultaneous 2nd | Total
Number analyzed (Participants) | 60 | 62 | 122
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 27 | 48
  >=65 years | 39 | 35 | 74
Age Continuous [Mean (Standard Deviation); unit: years] | 68.2 (14.1) | 66.1 (12.0) | 67.1 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 10 | 26
  Male | 44 | 52 | 96
Region of Enrollment [Number; unit: participants]
  United States | 58 | 59 | 117
  Switzerland | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Classified as "Not Worsened" for Changes in the Minnesota Living With Heart Failure Questionnaire and Six-minute Walk Distance Between Periods of Optimized and Simultaneous Biventricular Pacing
Description: The purpose is to evaluate the effectiveness of optimized pacing (OPT) compared to simultaneous pacing (SIM). The hypothesis is evaluated based on a responder classification. Subjects are classified "not worsened" if after 30 days of OPT the quality of life (QOL) score is no more than 10 points higher and the six-minute walk distance is no more than 35 meters lower than after 30 days of SIM. The Minnesota Living with Heart Failure questionnaire, a 21 question patient-completed survey, was used for QOL. Each question had a possible score of 0 (best) to 5 (worst), for a total of 0 to 105.
Time Frame: 60 days after enrollment
Population: Study utilized an intention-to-treat analysis. 111 out of 122 enrolled subjects completed the primary endpoint follow-up. 106 of these subjects met analysis criteria based on paired quality of life and six-minute walk data at the one and two month visits. Subjects not included in analysis either withdrew consent or had incomplete study measures.
Measure: Number; unit: Percent of Subjects
Groups:
- Total Subjects: Total subjects enrolled in study.
Arm/Group | Simultaneous 1st, Optimized 2nd | Optimized 1st, Simultaneous 2nd | Total Subjects
Number analyzed (Participants) | 51 | 55 | 106
Percent of Subjects | 65 | 62 | 63
Statistical Analysis 1: Comparison: Total Subjects; Efficacy was assessed in a non-inferiority, responder classification design where the proportion of total subjects classified as "not worsened" after changing from optimized to simultaneous biventricular pacing was compared to an objective performance criteria. An effect of gender analysis was performed on the primary efficacy endpoint to compare the proportion of males and females classified as "not worsened" after changing from optimized to simultaneous biventricular pacing; Test type: Non-Inferiority or Equivalence — The non-inferiority hypothesis utilized an objective performance criteria of 63% with a clinically significant difference of 12%. For the non-inferiority hypothesis, the one-sided Type I error was set to 0.05 and the statistical power was set to 80%; Non-inferiority comparison; Objective Performance Criteria = 63, 95% CI 1-sided [lower limit 54.8]

2. Primary Outcome: Percent of Subjects That Did Not Experience an Adverse Event That Require Additional Invasive Intervention to Resolve, Specifically Related to the Interventricular Delay Feature of the Lumax HF-T Heart Failure Device
Description: The purpose of primary endpoint two is to evaluate adverse events that require additional invasive intervention to resolve, specifically those events that are directly related to the interventricular delay feature of the Lumax HF-T heart failure device. These adverse events include any software issues related to the programming of the interventricular delay or any event that occurs after optimization of the interventricular delay and that can be directly attributed to the use of the feature.
Time Frame: 60 days after enrollment
Measure: Number; unit: Percent of Subjects
Arm/Group | Simultaneous 1st, Optimized 2nd | Optimized 1st, Simultaneous 2nd | Total Subjects
Number analyzed (Participants) | 60 | 62 | 122
Percent of Subjects | 100 | 100 | 100
Statistical Analysis 1: Comparison: Total Subjects; Safety will be evaluated in a non-inferiority format. The null hypothesis is the percent of subjects that did not experience an adverse event with an active interventricular delay feature at two months is inferior to 90% with a clinically significant difference of 10%; Test type: Non-Inferiority or Equivalence — The non-inferiority hypothesis has a one-sided Type I error of 0.05 with an 80% statistical power; Non-inferiority comparison; Objective Performance Criteria = 100, 95% CI 1-sided [lower limit 97.6]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected at each study visit until the final study visit at 6 months post enrollment.
Arm/Group | Simultaneous 1st, Optimized 2nd | Optimized 1st, Simultaneous 2nd | Total Subjects
Serious Adverse Events (participants affected / at risk) | 3/60 | 5/62 | 8/122
Other Adverse Events (participants affected / at risk) | 7/60 | 14/62 | 21/122
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Simultaneous 1st, Optimized 2nd (N=60) | Optimized 1st, Simultaneous 2nd (N=62) | Total Subjects (N=122)
Atrial arrhythmia requring invasive intervention to resolve (Cardiac disorders) | 1 (1) | 1 (1) | 2 (2)
Ventricular arrhythmia requiring invasive intervention to resolve (Cardiac disorders) | 0 (0) | 2 (2) | 2 (2)
Non-heart failure cardiac symptoms requiring invasive intervention to resolve (Cardiac disorders) | 1 (1) | 1 (1) | 2 (2)
Other cardiac condition requiring invasive intervention to resolve (Cardiac disorders) | 1 (1) | 3 (4) | 4 (5)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Simultaneous 1st, Optimized 2nd (N=60) | Optimized 1st, Simultaneous 2nd (N=62) | Total Subjects (N=122)
Worsening heart failure (Cardiac disorders) | 4 (4) | 8 (9) | 12 (13)
Other cardiac symptom (Cardiac disorders) | 3 (3) | 7 (8) | 10 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No